CLINICAL TRIAL: NCT00523068
Title: Randomized Pilot Study on the Treatment of Mixed Urinary Incontinence: Pharmacological Treatment (Tolterodine SR) vs Surgery With Tension Free Vaginal Tape
Brief Title: Pharmacological vs Surgical Treatment for Mixed Incontinence
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: it stopped at a regulatory stage
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/s0501/26
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Mixed Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge
Keywords: overactive bladder; stress urinary incontinence; detrusor overactivity; urodynamics
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tension Free Vaginal Tape
  Interventions: Procedure: tension free vaginal tape
- 2 (Active Comparator): Tolterodine tartrate 4mg
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Tolterodine
  Other Names: detrusitol XL
  Arms: 2
Procedure: tension free vaginal tape
  Arms: 1

SUMMARY:
In patients with symptoms of mixed incontinence (loss of urine associated with coughing/sneezing/laughing, and loss of urine associated with the strong urge to void), is surgical treatment with tension free vaginal tape or pharmacological treatment with tolterodine more effective? What are the parameters predictive of success or failure with either forms of treatment? What are the parameters predictive of the necessity for further treatment after primary treatment?

Patients will be randomised to having surgical or pharmacological treatment for their mixed incontinence symptoms. They will be assessed subjectively and objectively pre-treatment and after treatment at intervals up to 3 months.

DETAILED DESCRIPTION:
The aim of the study is to compare the efficacy and effect on the patient subsequent to pharmacological treatment with single dose tolterodine compared to surgical treatment with TVT in patients with urodynamically demonstrated mixed urinary incontinence, but with prevailing symptoms of stress incontinence. Secondary aims are the identification of parameters predictive of success or failure for the two treatments (echography, duration of the symptoms) and the necessity for further treatment after the primary therapy. The primary objective is to reduce the number of incontinence episodes after treatment with either modality.

The design will be randomisation of 40 patients, with 20 in the surgical group and 20 in the pharmacological treatment group. The patients must be female and aged between 35 and 70. They should not be intending to fall pregnant and be capable of completing a questionnaire about their incontinence symptoms and quality of life, a diary of their incontinence episodes and account of the passing of their urine, as well as be able to give informed consent to participate in the study.

The study will last for approximately 12 months and will consist of 5 visits. At the first visit, the patient will be seen to verify their suitability for admission into the study, have baseline blood tests, and urine analysis, as well as urodynamic assessment. They will also be given a diary to fill out an account of their urine passing which they will be asked to complete for the course of 3 days prior to their next appointment.

At the second appointment, the patient's diary will be collected and reviewed, a quality of life questionnaire will be completed, as well as an ultrasound scan performed to assess the thickness of the wall of their bladder. The patients will then be randomised into the pharmacological and surgical groups. Those in the surgical group will be put onto the waiting list for TVT (which they will have within 2 weeks of the second appointment), or commence treatment with tolterodine.

4 weeks after either treatment the patients are seen again and their symptoms are assessed and a second diary of the urinary behaviour (completed by the patient for the week prior to this visit) will be reviewed.

On the final visit, which will be after 12 weeks of treatment, the patients undergo urodynamic testing, diary assessment, symptom assessment, a quality of life questionnaire is completed and an appraisal of the patient's satisfaction with their treatment is collected. The discussion of need for any further treatment will take place and at this stage the patient may then have their treatment changed to either the tolterodine or surgery depending on their symptoms. These patients will then be finally seen after six months to review their progress.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female as this is a urogynaecology study.
2. An age of between 35 and 70 years. This takes into account that incontinence tends to prevail in women with advancing years. Younger women may be planning to start a family which precludes them from participating.
3. Clinical urodynamic evidence of mixed incontinence with prevalence of symptoms of stress incontinence assessed by means of a specific questionnaire and visual analog scale (VAS). The study is assessing the treatment of mixed incontinence and the patients will have to have evidence of this which is provided by their symptoms.
4. Candidates for corrective surgery of the component of sphincter defect with Ba < - 1 according to the International Continence Society (ICS) classification of genital prolapse.
5. Patients capable of filling in the micturition diary, the VAS, and the pathology specific quality of life questionnaire, the Kings Health Questionnaire. These form part of the continuing assessment of effectiveness of treatment.
6. Patients capable of understanding and signing an informed written consent form for participating in the trial. If patients are unable to give their consent for the procedures and investigations they cannot be ethically recruited.
7. Patients who accept not to give birth vaginally in the future, so as not to jeopardize the results of the surgical operation.

Exclusion Criteria:

1. Contraindications for using anti-cholinergic agents (urinary retention, uncontrolled narrow-angle glaucoma, myasthenia gravis, severe ulcerative colitis, toxic megacolon). Anticholinergics form one group of the patients and inability to take these drugs therefore precludes them from participating.
2. Ascertained hypersensitivity to tolterodine or any of the excipients. For the above reason.
3. Presence of pathologies or conditions that in the Investigator's opinion make the patient unsuitable for inclusion.
4. Patients with urinary tract infections (UTI) during the run-in period.
5. Patients with recurrent urinary tract infections (> 5 in the past 12 months).
6. Patients with diagnosed interstitial cystitis.

   These compromise the results obtained.
7. Patients with haematuria of uncertain origin. These patients need urgent investigation of these signs with procedures that are not included in the study.
8. Patients on treatment with anti-cholinergic agents of other drugs acting on detrusor instability. This will compromise the results of the study if for example these patients are randomised into the surgical group.
9. Patients on treatment with oestrogens, unless the therapy was commenced at least 2 months prior to inclusion in the study and follows a constant dosage.
10. Patients on diuretics. This affect their urinary behaviour.
11. Patients on concomitant treatment with potent CYP 34A inhibitors, such as macrolide antibiotics or antimycotic agents.
12. Patients who have undergone previous surgery on the distal urinary tract (with the exception of hysterectomy).
13. Patients who do not have adequate contraceptive cover or patients who are breast-feeding. For reasons of avoiding pregnancy during the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Estimated); Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
improvement in subjective and objective measures of urinary incontinence | 3 months

SECONDARY OUTCOMES:
assessment of pre-treatment predictors of success or failure of treatment | 3 months
assessment of pre-treatment predictors of requirement for alternative treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Khullar, Study Director — Imperial College London
Locations (1):
- Demetri C Panayi, London, United Kingdom